CLINICAL TRIAL: NCT01710046
Title: An Exploratory Phase 2a, Randomized, Double-blind, Placebo-controlled, Multicenter Study To Assess Mechanism Of Action (Moa) Of Cp-690,550 In The Skin When Administered Orally At 10 Mg Twice Daily (Bid) For 12 Weeks In Subjects With Moderate To Severe Chronic Plaque Psoriasis
Brief Title: Study Of The Mechanism Of Action Of CP-690,550 In The Skin Of Subjects With Moderate To Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3921147
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Results first posted 2015-04-13 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-03

CONDITIONS: Plaque Psoriasis
Keywords: plaque psoriasis; tofacitinib; biopsy; Janus Kinase; randomized placebo controlled clinical trial; psoriasis vulgaris
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental)
  Interventions: Drug: (CP-6890,550) Tofacitinib; Drug: Placebo
- Cohort 2 (Experimental)
  Interventions: Drug: (CP-690,550) Tofacitinib; Drug: Placebo

INTERVENTIONS:
Drug: (CP-6890,550) Tofacitinib — 2 x 5 mg oral capsules taken twice daily (every 12 hours) for 12 consecutive weeks
  Arms: Cohort 1
Drug: Placebo — 2 matching oral capsules taken twice daily (every 12 hours) for 12 consecutive weeks
  Arms: Cohort 1
Drug: (CP-690,550) Tofacitinib — 2 x 5 mg oral capsules taken twice daily (every 12 hours) for 12 weeks
  Arms: Cohort 2
Drug: Placebo — 2 matching oral capsules taken twice daily (every 12 hours) for 12 consecutive weeks
  Arms: Cohort 2

SUMMARY:
There are cells in the skin and blood of humans with chronic moderate to severe plaque psoriasis with specific activities that may determine the effectiveness of treatment. These activities may be described by obtaining samples of skin and blood and analyzing them using a variety of tests.

DETAILED DESCRIPTION:
The final subject in Cohort 1 completed the study on 19-Nov-2013 (LSLV date). Because the study analyses were novel and exploratory, they required extensive analyses by study team and external experts. As a result of this analysis it was determined on 21-July-2014 that the data from Cohort 1 were sufficiently definitive and that enrollment of Cohort 2 would not be justified. Since this decision resulted in the LSLV for Cohort 1 becoming the LSLV for the study, the full data analysis and reporting is not projected to be complete within 12 Months of LSLV. The final analysis and final reporting is planned to be completed on 18-Feb-2015. Results for this data are anticipated to be released in April 2015.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age with a diagnosis of chronic moderate to severe plaque psoriasis for at least 12 months; in generally good health; on stable dose of non-prohibited medications; able to stop current psoriasis therapy (systemic or topical) for several weeks prior to and during study participation.

Exclusion Criteria:

* Serious underlying disease including viral disorders such as hepatitis or HIV or skin condition that would interfere with skin biopsies or evaluation of psoriasis; conditions that could interfere with drug absorption after oral administration; history of malignancy or auto-immune disease.
* Use of oral or injected corticosteroids (steroids).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Dermatology Research Associates, Los Angeles, California
  - Olympian Clinical Research, Tampa, Florida
  - Menter Dermatology Research Institute, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas

REFERENCES:
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Krueger J, Clark JD, Suarez-Farinas M, Fuentes-Duculan J, Cueto I, Wang CQ, Tan H, Wolk R, Rottinghaus ST, Whitley MZ, Valdez H, von Schack D, O'Neil SP, Reddy PS, Tatulych S; A3921147 Study Investigators. Tofacitinib attenuates pathologic immune pathways in patients with psoriasis: A randomized phase 2 study. J Allergy Clin Immunol. 2016 Apr;137(4):1079-1090. doi: 10.1016/j.jaci.2015.12.1318. PMID 27059729
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921147&StudyName=Study%20Of%20The%20Mechanism%20Of%20Action%20Of%20CP-690%2C550%20In%20The%20Skin%20Of%20Subjects%20With%20Moderate%20To%20Severe%20Chronic%20Plaque%20Psoriasis

RESULTS

PARTICIPANT FLOW:
Groups:
- Tofacitinib 10 Milligrams (mg) Twice Daily (BID): Participants received tofacitinib tablets, 10 mg, orally, BID for 12 weeks.
- Placebo: Participants received matching placebo tablets, orally, BID for 12 weeks.
Period: Overall Study
Arm/Group | Tofacitinib 10 Milligrams (mg) Twice Daily (BID) | Placebo
Started | 9 | 3
Completed | 8 | 3
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tofacitinib 10 mg BID: Participants received tofacitinib tablets, 10 mg, orally, BID for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Tofacitinib 10 mg BID | Placebo | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.2 (11.3) | 46.7 (21.5) | 45.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 7 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a 75% Reduction in the Psoriasis Area and Severity Index (PASI75) at Week 12
Description: Combined assessment of lesion severity and area affected into single score; range equals (=) 0 (no disease) to 72 (maximal disease). Body divided into 4 sections=head, upper/lower limbs, trunk; each area scored by itself and scores combined for final PASI. For each section percent area of skin involved was estimated: 0 (0%) to 6 (90-100%) and severity estimated by clinical signs of erythema, induration, scaling; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final PASI=sum of severity parameters for each section*area score*weighing factor (head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4) summed over all sections.
Time Frame: Week 12
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 8 | 3
percentage of participants | 62.50 | 33.33

2. Primary Outcome: Percentage of Participants Achieving a Physician's Global Assessment (PGA) Response of "Clear" or "Almost Clear" at Week 12
Description: PGA psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration and scaling across all psoriatic lesions. PGA of Psoriasis scale ranges from 0 (no psoriasis) to 4 (severe disease). â€˜Clearâ€™ and â€œAlmost clearâ€™ includes all participants who were scored as a 0 or 1.
Time Frame: Week 12
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 8 | 3
percentage of participants | 50.00 | 33.33

3. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Score by Visit
Description: Combined assessment of lesion severity and area affected into single score. Body was divided into 4 sections: head, arms, trunk, legs. For each section, percent area of skin involved was estimated: 0=0% to 6=90â€"100%. Severity was estimated by clinical signs: erythema, induration, desquamation; scale: 0= none to 4= maximum. Final PASI = sum of severity parameters for each section*area score*weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4) summed over all sections; total possible score range: 0= no disease to 72= maximal disease.
Time Frame: Baseline and Weeks 1, 2, 4, and 12
Population: FAS; n (number) =number of participants with nonmissing observations at the specified visit.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 9 | 3
units on a scale
  Baseline (n=9,3) | 21.91 (2.86) | 23.33 (5.67)
  Week 1 (n=9,3) | 17.81 (3.10) | 15.53 (6.60)
  Week 2 (n=9,3) | 13.84 (2.71) | 13.13 (6.27)
  Week 4 (n=9,3) | 11.72 (3.51) | 13.37 (6.05)
  Week 12 (n=8,3) | 5.80 (1.80) | 13.40 (6.12)

4. Secondary Outcome: Change From Baseline in PASI by Visit
Description: as for outcome 3
Time Frame: Weeks 1, 2, 4 and 12
Population: Because Cohort 2 of the study was not conducted and Cohort 1 had a limited number of participants, the analyses were simplified and this analysis was not performed.
Arm/Group | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percent Change From Baseline in PASI by Visit
Description: Combined assessment of lesion severity and area affected into single score. Body was divided into 4 sections: head, arms, trunk, legs. For each section, percent area of skin involved was estimated: 0= 0% to 6= 90â€"100%. Severity was estimated by clinical signs: erythema, induration, desquamation; scale: 0= none to 4= maximum. Final PASI = sum of severity parameters for each section*area score*weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4) summed over all sections; total possible score range: 0= no disease to 72= maximal disease.
Time Frame: Weeks 1, 2, 4, and 12
Population: FAS; n=number of participants with nonmissing observations at the specified visit.
Measure: Mean (Standard Error); unit: percent change from baseline
Arm/Group | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 9 | 3
percent change from baseline
  Week 1 (n=9,3) | -18.38 (7.52) | -39.61 (19.97)
  Week 2 (n=9,3) | -36.95 (8.28) | -48.66 (20.28)
  Week 4 (n=9,3) | -47.39 (11.95) | -49.66 (19.41)
  Week 12 (n=8,3) | -71.78 (9.63) | -49.13 (19.67)

6. Secondary Outcome: Percentage of Participants Achieving a PASI75 Response at Weeks 1, 2, and 4
Description: Combined assessment of lesion severity and area affected into single score; range=0 (no disease) to 72 (maximal disease). Body divided into 4 sections=head, upper/lower limbs, trunk; each area scored by itself and scores combined for final PASI. For each section percent area of skin involved was estimated: 0 (0%) to 6 (90-100%) and severity estimated by clinical signs of erythema, induration, scaling; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final PASI=sum of severity parameters for each section*area score*weighing factor (head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4) summed over all sections.
Time Frame: Weeks 1, 2, and 4
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 9 | 3
percentage of participants
  Week 1 | 0.00 | 0.00
  Week 2 | 0.00 | 33.33
  Week 4 | 22.22 | 33.33

7. Secondary Outcome: Change From Baseline in PGA Score by Visit
Description: PGA psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. PGA of Psoriasis scale ranges from 0 (no psoriasis) to 4 (severe disease). The severity scores of 3 components (erythema, induration, and scaling) are averaged and rounded to the nearest whole number to determine the PGA score.
Time Frame: Weeks 1, 2, 4, and 12
Population: FAS; n=number of participants with nonmissing observations at the specified visit.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 9 | 3
units on a scale
  Week 1 (n=9,3) | -0.6 (0.2) | -0.7 (0.3)
  Week 2 (n=9,3) | -0.8 (0.2) | -1.0 (0.6)
  Week 4 (n=9,3) | -1.2 (0.3) | -1.0 (0.6)
  Week 12 (n=8,3) | -1.5 (0.3) | -1.0 (0.6)

8. Secondary Outcome: Percentage of Participants in Each PGA Category at Various Timepoints by Baseline Category
Time Frame: Baseline and Weeks 1, 2, 4, and 12
Population: as for outcome 4
Arm/Group | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percentage of Participants by PGA Response Category and Timepoint
Description: PGA psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration and scaling across all psoriatic lesions. PGA of Psoriasis scale ranges from 0 (no psoriasis) to 4 (severe disease). Response category scores: 0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe. The severity scores of 3 components (erythema, induration, and scaling) are averaged and rounded to the nearest whole number to determine the PGA score.
Time Frame: Baseline and Weeks 1, 2, 4, and 12
Population: FAS; n=number of participants with nonmissing observations at the specified visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 9 | 3
percentage of participants
  Baseline, Moderate (n=9,3) | 88.9 | 66.7
  Baseline, Severe (n=9,3) | 11.1 | 33.3
  Week 1, Mild (n=9,3) | 44.4 | 33.3
  Week 1, Moderate (n=9,3) | 55.6 | 66.7
  Week 2, Almost clear (n=9,3) | 11.1 | 33.3
  Week 2, Mild (n=9,3) | 44.4 | 0
  Week 2, Moderate (n=9,3) | 44.4 | 66.7
  Week 4, Almost clear (n=9,3) | 44.4 | 33.3
  Week 4, Mild (n=9,3) | 22.2 | 0
  Week 4, Moderate (n=9,3) | 33.3 | 66.7
  Week 12, Almost clear (n=8,3) | 50.0 | 33.3
  Week 12, Mild (n=8,3) | 37.5 | 0
  Week 12, Moderate (n=8,3) | 12.5 | 66.7

10. Secondary Outcome: Body Surface Area (BSA)
Description: Assessment of BSA with psoriasis was performed separately for 4 body regions: head and neck, upper limbs, trunk (including axillae and groin), and lower limbs (including buttocks). The percent surface area with psoriasis was estimated by means of the handprint method, where the full palmar hand of the participant (ie, the participant's fully extended palm, fingers and thumb together) represents approximately 1% of the total BSA. The number of handprints of psoriatic skin in a body region can be used to determine the extent (%) to which a body regions is involved with psoriasis. In each body region, the percent body region surface area with psoriasis is multiplied by the Body Region Weighting (head and neck=10%, upper limbs=5%, trunk [including axillae and groin]=3.33% and lower limbs [including buttocks]=2.5%). BSA (%)=0.1Sh + 0.2Sh+0.3St+0.4Sl, where S=body region suface area with psoriasis: h=head; u=upper limbs; t=trunk; l=lower limbs.
Time Frame: Baseline and Weeks 1, 2, 4, and 12
Population: FAS; n=number of participants with nonmissing observations at the specified visit.
Measure: Mean (Standard Error); unit: % BSA
Arm/Group | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 9 | 3
% BSA
  Baseline (n=9,3) | 34.16 (8.12) | 30.50 (10.87)
  Week 1 (n=9,3) | 31.20 (7.35) | 24.83 (10.43)
  Week 2 (n=9,3) | 24.20 (5.38) | 24.67 (10.59)
  Week 4 (n=9,3) | 19.03 (4.70) | 23.33 (10.43)
  Week 12 (n=8,3) | 7.35 (3.10) | 23.03 (10.50)

11. Secondary Outcome: Change From Baseline in BSA
Description: as for outcome 10
Time Frame: Weeks 1, 2, 4, and 12
Population: as for outcome 4
Arm/Group | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percent Change From Baseline in BSA
Description: as for outcome 10
Time Frame: Weeks 1, 2, 4, and 12
Population: FAS; n=number of participants with nonmissing observations at the specified visit.
Measure: Mean (Standard Error); unit: percent change from baseline
Arm/Group | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 9 | 3
percent change from baseline
  Week 1 (n=9,3) | -6.87 (4.97) | -27.80 (17.46)
  Week 2 (n=9,3) | -22.51 (7.14) | -29.47 (19.01)
  Week 4 (n=9,3) | -35.13 (10.45) | -34.93 (21.80)
  Week 12 (n=8,3) | -77.40 (11.98) | -37.26 (21.53)

13. Secondary Outcome: Itch Severity Item (ISI) Score by Visit
Description: The severity of itch (pruritus) due to psoriasis was assessed using the ISI, a single-item, horizontal numeric rating scale. Participants were asked to rate "your worst itching due to psoriasis over the past 24 hours" on a numeric rating scale anchored by the terms "No itching" (0) and "Worst possible itching" (10) at the ends. the baseline is defined as the average of all available diary entries before Baseline/Day 1 and the in-clinic measurement on Baseline/day 1. Week 1 is the mean of daily values of study days 2 to 8 and Week 2 is the mean of daily values of study days 9 to 15.
Time Frame: Baseline and Weeks 1, 2, 4, and 12
Population: FAS; n=number of participants with nonmissing observations at the specified visit.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 9 | 3
units on a scale
  Baseline (n=9,3) | 6.35 (0.89) | 3.46 (1.94)
  Week 1 (n=9,3) | 3.81 (0.97) | 3.90 (1.73)
  Week 2 (n=9,3) | 2.45 (0.91) | 1.99 (0.73)
  Week 4 (n=9,3) | 1.22 (0.57) | 2.67 (1.20)
  Week 12 (n=8,3) | 0.75 (0.62) | 6.00 (1.53)

14. Secondary Outcome: Change From Baseline in ISI by Visit
Description: ISI, a single-item, horizontal numeric rating scale. Participants were asked to rate "your worst itching due to psoriasis over the past 24 hours" on a numeric rating scale anchored by the terms "No itching" (0) and "Worst possible itching" (10) at the ends. The baseline is defined as the average of all available diary entries before Baseline/Day 1 and the in-clinic measurement on Baseline/Day 1. Week 1 is the mean of daily values of study days 2 to 8 and Week 2 is the mean of daily values of study days 9 to 15. A negative value indicates an improvement.
Time Frame: Weeks 1, 2, 4 and 12
Population: FAS; n=number of participants with nonmissing observations at the specified visit.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 9 | 3
units on a scale
  Week 1 (n=9,3) | -2.55 (0.59) | 0.45 (0.52)
  Week 2 (n=9,3) | -3.90 (0.67) | -1.47 (1.31)
  Week 4 (n=9,3) | -5.13 (0.77) | -0.79 (2.35)
  Week 12 (n=8,3) | -5.96 (0.99) | 2.54 (2.61)

15. Secondary Outcome: Target Plaque Severity Score (TPSS) by Visit
Description: Target lesions were selected at baseline and followed for the duration of the study. Each target lesion was scored by the investigator on severity of erythema, induration, and scaling according to a 5-point (0 to 4) severity scale with a maximum sum score for a plaque of 12. The TPSS was calculated as the sum of the scores for erythema, induration, and scaling; the score can vary in increments of 1 unit from 0 to 12.
Time Frame: Baseline and Weeks 1, 2, 4, and 12
Population: FAS; n=number of participants with nonmissing observations at the specified visit.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 9 | 3
score on a scale
  Baseline (n=9,3) | 8.7 (0.6) | 8.3 (0.3)
  Week 1 (n=9,3) | 7.1 (0.7) | 7.0 (1.2)
  Week 2 (n=9,3) | 6.0 (0.7) | 6.7 (1.2)
  Week 4 (n=9,3) | 4.6 (1.1) | 6.7 (1.9)
  Week 12 (n=8,3) | 2.8 (1.3) | 6.0 (1.7)

16. Secondary Outcome: Percent Change From Baseline in TPSS by Visit
Description: Target lesions were selected at baseline and followed for the duration of the study. Each target lesion was scored by the investigator on severity of erythema, induration, and scaling according to a 5-point (0 to 4) severity scale with a maximum sum score for a plaque of 12. The TPSS was calculated as the sum of the scores for erythema, induration, and scaling; the score can vary in increments of 1 unit from 0 to 12. A negative value indicated improvment.
Time Frame: Weeks 1, 2, 4, and 12
Population: FAS; n=number of participants with nonmissing observations at the specified visit.
Measure: Mean (Standard Error); unit: percent change from baseline
Arm/Group | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 9 | 3
percent change from baseline
  Week 1 (n=9,3) | -16.69 (7.72) | -16.67 (11.02)
  Week 2 (n=9,3) | -29.78 (8.39) | -20.83 (11.02)
  Week 4 (n=9,3) | -47.55 (12.40) | -20.83 (20.83)
  Week 12 (n=8,3) | -67.28 (15.17) | -29.17 (18.16)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from the time of informed consent through and including 28 calendar days after the last administration of the investigational product.
Description: The same event may appear as both an AE and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Tofacitinib 10 mg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/3
Other Adverse Events (participants affected / at risk) | 2/9 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 10 mg BID (N=9) | Placebo (N=3)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 10 mg BID (N=9) | Placebo (N=3)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Gravitational oedema (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No